CLINICAL TRIAL: NCT01513343
Title: Promoting The Self-Regulation Of Energy Intake In Latino Preschoolers: A Family Focused Obesity Prevention Program
Brief Title: Promoting The Self-Regulation Of Energy Intake
Acronym: SEEDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Washington State University (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Sheryl Hughes, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USDA 2011-68001-30009; H-28013 (Other: Baylor College of Medicine)
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent and child classes (prevention group) (Experimental): Parent and child groups focused on self-regulation of eating
  Interventions: Behavioral: Parent and child groups focused on self-regulation of eating
- Treatment as usual (control group) (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Parent and child groups focused on self-regulation of eating
  Arms: Parent and child classes (prevention group)

SUMMARY:
The goal of this study is to develop and test the efficacy of a scientifically-based, culturally competent seven-session parent directed, obesity prevention program focused on parental feeding strategies that support young children's self-regulation of intake.

DETAILED DESCRIPTION:
The intervention program was developed and piloted. Expected outcomes: At the end of the intervention program, it is expected that parents in the intervention group will: 1) use more child-centered (e.g., repeated presentation of new foods, involvement in food preparation) and less parent-centered feeding directives; 2) be less likely to show an indulgent and more likely to show an authoritative feeding style (feeding responsiveness); 3) show lower scores on restriction and pressure to eat and higher scores on monitoring; and 4) demonstrate higher levels of food knowledge (e.g., best feeding practices, reduced feeding misconceptions). Children in the intervention group are expected to: 1) show more willingness to try new foods, and 2) show increased self-regulation of energy intake. At the end of the interventions, children are expected to show greater consumption of fruits and vegetables (including consuming a wider variety of fruits and vegetables). All effects are expected to continue through the 6- and 12-month follow-ups, although the effects sizes will diminish. Although we do not expect effects on BMI after 6 weeks, we expect to see decreases in children's BMI percentiles by the 6- and 12-month follow-ups for the intervention group-especially for the top 25% of the BMI percentile range. No parental BMI effects are expected.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children attend Head Start with the sample of children equally split on gender and ethnicity,
* with representation from ages 3 to 6 years.

Exclusion Criteria:

* Parents and children who have any kind of food allergies or diabetes or are on special diets will be excluded from the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2014-08; Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O Hughes, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Thomas G. Power, Pullman, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parent/child dyads were recruited in 2014-2016 from Head Start centers in Houston, TX, and child care centers serving families with low incomes in Pasco, WA. The Pasco centers were similar to Head Start in that they provided free services and support for families with low incomes. The goal of these centers was to ensure that all children enter kindergarten ready to succeed.
Pre-assignment Details: No significant events occurred in this study after participant enrollment.
Groups:
- Treatment as Usual (Control Group): Treatment as usual, parents and children did not receive any treatment as the control group.
Period: Group Allocation
Arm/Group | Parent and Child Classes (Prevention Group) | Treatment as Usual (Control Group)
Started (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 136 | 119
Completed (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 128 | 119
Not Completed | 8 | 0
Not completed — Dropped out after randomization, did not attend any lessons, included in analyses as intent-to-treat | 8 | 0
Period: Post Data Collection
Arm/Group | Parent and Child Classes (Prevention Group) | Treatment as Usual (Control Group)
Started (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 136 | 119
Completed (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 119 | 95
Not Completed | 17 | 24
Not completed — Dropped/withdrew from study | 7 | 1
Not completed — Lost to Follow-up | 10 | 23
Period: 6-month Follow-up
Arm/Group | Parent and Child Classes (Prevention Group) | Treatment as Usual (Control Group)
Started (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 119 | 95
Completed (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 91 | 78
Not Completed | 28 | 17
Not completed — Lost to Follow-up | 28 | 17
Period: 12-month Follow-up
Arm/Group | Parent and Child Classes (Prevention Group) | Treatment as Usual (Control Group)
Started (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 91 | 78
Completed (Numbers reported reflect parent/child dyads; there are 2 unique participants within each dyad.) | 81 | 75
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 10 | 3

BASELINE CHARACTERISTICS:
Population: A total of 255 parent/child dyads participated in the study (255 parents and their children). We report age, gender, and ethnicity for children and parents separately, thus there are 2 entries each for age, gender, and ethnicity (one for children and one for parents).
  All analyses were intention-to-treat analyses. Specifically, data from parents and children were analyzed on the basis of the condition to which they were initially assigned, regardless of the number of classes they attended.
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent and Child Classes (Prevention Group) | Treatment as Usual (Control Group) | Total
Number analyzed (Participants) | 136 | 119 | 255
Age, Continuous [Mean (Standard Deviation); unit: months] — Child age in months Population: Data on child age are missing for 1 child in the prevention group and 2 children in the control group.
  months
    number analyzed (Participants) | 135 | 117 | 252
    (all) | 56.28 (7.11) | 54.61 (6.84) | 55.40 (7.02)
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent age in years Population: Data on parent age are missing for 4 parents in the prevention group and 3 parents in the control group.
  years
    number analyzed (Participants) | 132 | 116 | 248
    (all) | 33.95 (7.12) | 32.53 (6.92) | 33.29 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants] — Parent-report of child sex
  Participants
    Female | 73 | 53 | 126
    Male | 63 | 66 | 129
Sex: Female, Male [Count of Participants; unit: Participants] — Parent self-report of sex
  Participants
    Female | 136 | 119 | 255
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent-report of child ethnicity
  Participants
    Hispanic or Latino | 136 | 119 | 255
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent self-report of ethnicity
  Participants
    Hispanic or Latino | 136 | 119 | 255
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Parent/child dyad] — Data were collected from both parents and their children and data are reported as family unit, i.e., parent/child dyads. Data were collected from dyads in Houston, TX and Pasco, WA.
  Parent/child dyad
    United States | 136 | 119 | 225
Children's BMI Percentiles [Count of Participants; unit: Participants] — Measured child height and weight data were collected. Two height and weight measures were averaged for each child. Age- and gender-specific BMI z-scores for each child were calculated. Children were classified into healthy weight (5th to <85th percentile), overweight (≥85th to <95th percentile), and obese (≥95th percentile) according to Centers for Disease Control and Prevention standards. Population: Child height and weight data were not available for 2 participants in the "parent and child classes" group and 2 participants in the "treatment as usual" group.
  Participants
    number analyzed (Participants) | 134 | 117 | 251
    Healthy weight (<85th percentile) | 78 | 79 | 157
    Overweight (85th to 95th percentile) | 27 | 21 | 48
    Obese (≥95th percentile) | 29 | 17 | 46

OUTCOME MEASURES:

1. Primary Outcome: Children's BMI Percentiles
Description: Measured child height and weight data were collected. Two height and weight measures were averaged for each child. Age- and gender-specific BMI z-scores for each child were calculated. Children were classified into healthy weight (5th to <85th percentile), overweight (≥85th to <95th percentile), and obese (≥95th percentile) according to Centers for Disease Control and Prevention standards.
Time Frame: 12-month follow-up
Population: Prevention group: 76 children assessed at 12-months.
  Treatment as usual control group: 71 children assessed at 12-months.
Measure: Count of Participants; unit: Participants
Groups:
- Prevention Group: Focused on self-regulation of eating
- Treatment as Usual Control Group: Treatment as usual control group did not receive any treatment
Arm/Group | Prevention Group | Treatment as Usual Control Group
Number analyzed (Participants) | 76 | 71
Participants
  Healthy weight (<85th percentile) | 49 | 41
  Overweight (85th to 95th percentile) | 15 | 18
  Obese (≥95th percentile) | 12 | 12
Statistical Analysis 1: Comparison: Prevention Group vs Treatment as Usual Control Group; Test type: Superiority; p < 0.05, Regression, Logistic; Multinomial logistic regression examined program effects on child BMI categories, controlling for child sex, age (months), & BMI z-score at pretest

2. Secondary Outcome: Parental Feeding Behaviors
Description: Questionnaire data (parent-report). Subscale scores from the Food Parenting Inventory and Feeding Knowledge Questionnaire were used to measure secondary outcomes. All scales included response categories ranging from 1 to 5. Higher scores were considered better on the following subscales: repeated presentation of new foods; measured child portion sizes; child involvement in food preparation; feeding responsiveness; knowledge of best feeding practices; feeding efficacy. Lower scores were considered better on the subscale of feeding misconceptions.
Time Frame: 12-month follow-up
Population: Prevention group: 67 parents assessed at 12-months.
  Treatment as usual control group: 54 parents assessed at 12-months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Prevention Group: Group focused on self-regulation of eating
Arm/Group | Prevention Group | Treatment as Usual Control Group
Number analyzed (Participants) | 67 | 54
score on a scale
  repeated presentation of new foods: number analyzed (Participants) | 67 | 53
  repeated presentation of new foods | 3.5 [3.30 to 3.70] | 3.2 [3.02 to 3.44]
  measured child portion sizes: number analyzed (Participants) | 67 | 53
  measured child portion sizes | 3.1 [2.82 to 3.32] | 2.5 [2.23 to 2.74]
  child involvement in food preparation: number analyzed (Participants) | 67 | 53
  child involvement in food preparation | 2.9 [2.69 to 3.10] | 2.8 [2.54 to 2.96]
  feeding responsiveness: number analyzed (Participants) | 67 | 53
  feeding responsiveness | 3.8 [3.60 to 4.02] | 3.4 [3.18 to 3.62]
  knowledge of best feeding practices: number analyzed (Participants) | 65 | 54
  knowledge of best feeding practices | 4.1 [4.00 to 4.21] | 3.9 [3.81 to 4.02]
  feeding misconceptions: number analyzed (Participants) | 65 | 54
  feeding misconceptions | 3.0 [2.85 to 3.11] | 3.2 [3.10 to 4.02]
  feeding efficacy: number analyzed (Participants) | 65 | 54
  feeding efficacy | 4.2 [4.07 to 4.39] | 4.0 [3.81 to 4.13]
Statistical Analysis 1: Comparison: Prevention Group vs Treatment as Usual Control Group; Test type: Superiority; p < 0.05, Mixed Models Analysis — To control for type I errors, the critical P values for each assessment were determined with the unweighted Bonferroni method, dividing the critical value of P < 0.05 by the number of comparisons conducted for a given assessment

ADVERSE EVENTS:
Time Frame: Adverse events were monitored between August 2014 and December 2017.
Arm/Group | Prevention Group | Treatment as Usual Control Group
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/119
Other Adverse Events (participants affected / at risk) | 0/136 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT01513343/Prot_SAP_000.pdf